CLINICAL TRIAL: NCT03270436
Title: Diabetes Prevention Program Lifestyle Intervention in the Marshallese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 207034
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Comparison of two diabetes prevention program curricula in the Marshallese population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program (Experimental): The Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program (WORD DPP) is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length. The first 8 modules are intended to be delivered weekly. The last 8 modules are intended to be delivered every other week. Participants in the WORD DPP will be encouraged to maintain a daily weight, nutrition, physical activity and prayer log.
  Interventions: Behavioral: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program
- Partnership for Improving Lifestyle Intervention Diabetes Prevention Program (Experimental): The Partnership for Improving Lifestyle Intervention Diabetes Prevention Program (PILI DPP) is a family and community based diabetes prevention curriculum that teaches participants to engage their social support (family and community) to have a healthy weight, eat healthy, and be physically active. The PILI DPP includes 14 modules that are intended to be delivered over a 24 week period and each module approximately 90 minutes in length. The first 4 modules are intended to be delivered weekly. The last 10 modules are intended to be delivered every other week. Participants will be encouraged to track their weight, physical activity, and their nutrition in a log on a daily basis.
  Interventions: Behavioral: Partnership for Improving Lifestyle Intervention Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program — Faith based diabetes curriculum that teaches participants to connect faith and health.
  Arms: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program
Behavioral: Partnership for Improving Lifestyle Intervention Diabetes Prevention Program — Family and community based diabetes prevention curriculum that teaches participants to engage their social support to have a healthy weight.
  Arms: Partnership for Improving Lifestyle Intervention Diabetes Prevention Program

SUMMARY:
The investigators will conduct a comparative effectiveness cluster-randomized controlled trial (cRCT) of two Diabetes Prevention Program (DPP) lifestyle interventions: a faith-based intervention (Wholeness, Oneness, Righteousness, Deliverance [WORD] DPP); and a Pacific Islander adapted intervention (Partnership for Improving Lifestyle Interventions [PILI] DPP. Each intervention lasted 24 weeks and focused on the importance of healthy eating, being physically active, and maintaining a healthy weight. Eligible participants included overweight and obese Marshallese adults living in Arkansas and Oklahoma. The unit of randomization is at the church level. The primary outcome measure is body weight loss (from baseline weight). As selected by stakeholders, HbA1c, blood pressure, physical activity, and dietary intake will be evaluated as secondary outcome measures. Data collection will take place at baseline (pre-intervention), immediate post-intervention (6 months post-initiation of the intervention), and 6 months post-intervention (12 months post-initiation of the intervention).

DETAILED DESCRIPTION:
Background and Rationale

Disparities in type 2 diabetes, pre-diabetes, and obesity among the Marshallese and Pacific Islanders.

The Marshallese are a Pacific Islander population experiencing significant health disparities, with some of the highest documented rates of type 2 diabetes of any population group in the world. Our review of local, national, and international data sources found estimates of diabetes in the Marshallese population (those living in the US and in the Republic of the Marshall Islands) ranging from 20% to 50%, compared to 8.3% for the US population and 4% worldwide. While national prevalence data are limited, 23.7% of Pacific Islanders surveyed by the Centers for Disease Control and Prevention (CDC) in 2010 reported a diagnosis of type 2 diabetes, more than all other racial/ethnic groups. Our pilot research, which includes health screenings with the Marshallese community in northwest Arkansas (n=398), documented extremely high incidence of diabetes (38.4%) and pre-diabetes (32.6%). Our pilot data also revealed similar disparities in one of the strongest risk factors for diabetes-obesity-with 90% of Marshallese participants classified as overweight or obese. Thirty-two percent of those who had pre-diabetes were also overweight or obese. Further compounding these significant disparities in diabetes prevalence and related risk factors, research indicates that Pacific Islanders living in the US are less likely than other racial/ethnic groups to receive preventative or diagnostic treatment, or diabetes education.

Reducing disparities by reducing weight. Overweight/obesity is considered the strongest modifiable risk factor for type 2 diabetes, and even a modest reduction in weight (5-10%) can be clinically meaningful.

Specific aim. Our aim is to compare the effectiveness of achieving weight loss between two Diabetes Prevention Program (DPP) Lifestyle Interventions - the faith-based Wholeness, Oneness, Righteousness, Deliverance (WORD) DPP, and the Pacific Islander culturally-adapted Partnership for Improving Lifestyle Interventions (PILI) DPP - in the Marshallese population using a cluster randomized controlled trial (cRCT).

Study design. The study design is a comparative effectiveness cRCT conducted in church settings or other community setting convenient to the participant group. Churches were selected as the primary setting based on Marshallese stakeholder input.

Randomized participant assignment. Randomization will occur at the church cluster level, with 1:1 assignment of churches to each arm. Churches and community based participant groups will be blocked (i.e., grouped into similar units) according to geographic region and approximate number of adult church members. Randomization will be conducted by a biostatistician or designated investigator, who will have no interactions with potential participants and has no supervisory role with study staff responsible for recruiting, consent, and intervention process.

Recruitment and Consent

Church-based recruitment is specified by stakeholders as culturally appropriate and the community's preferred recruitment method. During recruitment, Marshallese study staff will give presentations and distribute study information in English and Marshallese. Those who express interest will complete an eligibility screener, to determine eligibility. All study information and consent materials will be provided in English and/or Marshallese based upon the participants' preferences. Eligible participants will be provided a copy of the consent to review, and participants will have the opportunity to ask questions, consent, and enroll in the study. The consent process will include providing information to the potential participants and the opportunity to have bilingual Marshallese staff answer questions regarding study participation. The consent document will be given to the participant, and the informed consent process will be documented in the participant's research record.

ELIGIBILITY:
Inclusion Criteria:

* Self reported Marshallese
* 18 years of age or older
* BMI greater than or equal to 25

Exclusion Criteria:

* A clinically significant medical condition likely to impact weight (cancer, HIV/AIDS, etc.)
* Currently pregnant or breastfeeding an infant who is 6 months old or younger
* Have any condition that makes it unlikely that the participant will be able to follow the protocol, such as terminal illness, plans to move out of the area within 6 months, an inability to finish the intervention, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McElfish PA, Felix HC, Bursac Z, Rowland B, Yeary KHK, Long CR, Selig JP, Kaholokula JK, Riklon S. A Cluster Randomized Controlled Trial Comparing Diabetes Prevention Program Interventions for Overweight/Obese Marshallese Adults. Inquiry. 2023 Jan-Dec;60:469580231152051. doi: 10.1177/00469580231152051. PMID 36799349
- [Derived] McElfish PA, Long CR, Kaholokula JK, Aitaoto N, Bursac Z, Capelle L, Laelan M, Bing WI, Riklon S, Rowland B, Ayers BL, Wilmoth RO, Langston KN, Schootman M, Selig JP, Yeary KHK. Design of a comparative effectiveness randomized controlled trial testing a faith-based Diabetes Prevention Program (WORD DPP) vs. a Pacific culturally adapted Diabetes Prevention Program (PILI DPP) for Marshallese in the United States. Medicine (Baltimore). 2018 May;97(19):e0677. doi: 10.1097/MD.0000000000010677. PMID 29742712

RESULTS

PARTICIPANT FLOW:
Groups:
- Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program: The Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program (WORD DPP) is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length. The first 8 modules are intended to be delivered weekly. The last 8 modules are intended to be delivered every other week. Participants in the WORD DPP will be encouraged to maintain a daily weight, nutrition, physical activity and prayer log.
  WORD DPP: Faith based diabetes curriculum that teaches participants to connect faith and health.
- Partnership for Improving Lifestyle Intervention Diabetes Prevention Program: The Partnership for Improving Lifestyle Intervention Diabetes Prevention Program (PILI DPP) is a family and community based diabetes prevention curriculum that teaches participants to engage their social support (family and community) to have a healthy weight, eat healthy, and be physically active. The PILI DPP includes 14 modules that are intended to be delivered over a 24 week period and each module approximately 90 minutes in length. The first 4 modules are intended to be delivered weekly. The last 10 modules are intended to be delivered every other week. Participants will be encouraged to track their weight, physical activity, and their nutrition in a log on a daily basis.
  PILI DPP: Family and community based diabetes prevention curriculum that teaches participants to engage their social support to have a healthy weight.
Period: Baseline
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Started | 213 | 167
Completed | 212 | 166
Not Completed | 1 | 1
Period: Immediate Post-Intervention
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Started (All enrolled participants were contacted to provide data at post-intervention whether or not they completed baseline data collection.) | 213 | 167
Completed | 172 | 111
Not Completed | 41 | 56
Period: 6 Months Post-Intervention
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Started (All enrolled participants were contacted to provide data at 6 months post-intervention whether or not they completed previous data collections.) | 213 | 167
Completed | 173 | 116
Not Completed | 40 | 51

BASELINE CHARACTERISTICS:
Population: The total number of participants providing data at baseline data collection.Two enrolled participants failed to provide data at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program | Total
Number analyzed (Participants) | 212 | 166 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (10.6) | 41.4 (12.8) | 42.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 97 | 214
  Male | 95 | 69 | 164
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 212 | 166 | 378
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 212 | 166 | 378
Weight (kg) [Mean (Standard Deviation); unit: kg] — Participant weight (without shoes) was measured in light clothing using a calibrated digital scale.
  kg | 85.4 (15.6) | 83.4 (14.3) | 84.4 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Body Weight (kg)
Description: Change in mean body weight (kg) from baseline to immediate post intervention and 6 months post-intervention. Participant weight (without shoes) was measured in light clothing using a calibrated digital scale at each time point.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: Kilograms
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
Kilograms
  Baseline | 86.44 (1.65) | 84.32 (1.80)
  Immediate post-intervention | 86.47 (1.72) | 84.40 (1.97)
  6 months post-intervention | 86.18 (1.84) | 83.80 (2.10)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.3599, linear mixed effects regression — The p-value above reflects results of between-arms analysis of change in mean weight from baseline to immediate post-intervention. Analyses do not include imputed values; Model includes group, time, g x t interaction, state, age, gender, marital status, employment, education, and accounts for clustering within churches
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.3207, linear mixed effects regression — The p-value above reflects results of between-arms analysis of change in mean weight from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Mean HbA1c (%)
Description: Change in mean HbA1c (NGSP %) from baseline to immediate post-intervention and 6 months post-intervention. A Siemens analyzer (point of care) was utilized to calculate HbA1c levels for each participant at each time point.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: Percent Glycated Hemoglobin
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
Percent Glycated Hemoglobin
  Baseline | 7.27 (0.30) | 7.66 (0.33)
  Immediate post-intervention | 7.32 (0.31) | 7.55 (0.36)
  6 months post-intervention | 7.25 (0.33) | 7.61 (0.38)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.5698, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in HbA1c from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.4106, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in HbA1c from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Mean Systolic Blood Pressure (mmHg)
Description: Change in mean systolic blood pressure (mmHg) from baseline to immediate post-intervention and 6 months post-intervention. Blood pressure was measured at each time point with a sphygmomanometer and stethoscope or digital blood pressure device, with participants seated and arm elevated.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
mmHg
  Baseline | 129.42 (2.39) | 128.20 (2.60)
  Immediate post-intervention | 126.83 (2.47) | 119.65 (2.82)
  6 months post-intervention | 120.75 (2.61) | 118.30 (2.96)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.0293, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in systolic blood pressure from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.4686, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in systolic blood pressure from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Mean Diastolic Blood Pressure (mmHg)
Description: Change in mean diastolic blood pressure (mmHg) from baseline to immediate post-intervention and 6 months post-intervention. Blood pressure was measured at each time point with a sphygmomanometer and stethoscope or digital blood pressure device, with participants seated and arm elevated.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
mmHg
  Baseline | 79.60 (1.12) | 78.33 (1.22)
  Immediate post-intervention | 78.50 (1.19) | 74.08 (1.38)
  6 months post-intervention | 76.41 (1.29) | 76.24 (1.49)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.0068, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in diastolic blood pressure from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.9181, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in diastolic blood pressure from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Sugar-sweetened Beverage Consumption
Description: Change in participants' sugar-sweetened beverage (SSB) consumption from baseline to immediate post-intervention and 6 months post-intervention. This self-report measure assessed participants' SSB consumption over the past 30 days using two questions from 'Module 14: Sugar Sweetened Beverages' of the Center for Disease Control and Prevention's Behavioral Risk Factor Surveillance System (BRFSS). Participants could respond in number of times per day, per week, or per month. Responses for each question were converted to number of times per day (i.e., self-reported times per week divided by 7 or self-reported times per month divided by 30), resulting in two measures: number times soda was consumed per day and number of times sugar-sweetened fruit drinks, sweet tea, and sports drinks were consumed per day. Per BRFSS guidelines, these two measures were added together to create a total daily SSB consumption rate.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: SSBs consumed per day
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
SSBs consumed per day
  Baseline | 1.65 (0.16) | 2.16 (0.17)
  Immediate post-intervention | 1.24 (0.17) | 1.36 (0.20)
  6 months post-intervention | 1.18 (0.17) | 1.40 (0.20)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.5984, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in sugar-sweetened beverages consumed per day from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.3376, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in sugar-sweetened beverages consumed per day from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Change in Fruit and Vegetable Consumption
Description: Change in participants' fruit and vegetable consumption from baseline to immediate post-intervention and 6 months post-intervention. This self-report measure assessed participants' fruit and vegetable consumption over the past three months using three items adapted from: Shannon J, Kristal AR, Curry SJ, Beresford SA. Application of a behavioral approach to measuring dietary change: the fat- and fiber-related diet behavior questionnaire. Cancer Epidemiol Biomarkers Prev. 1997;6(5):355-361. Each of the three items was scored as Often=2; Sometimes=1; Never=0. Items were summed to create a scale score, giving a possible range of scores of 0-6, with higher scores indicating more frequent consumption of fruits and vegetables.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: scale score
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
scale score
  Baseline | 3.59 (0.15) | 3.70 (0.16)
  Immediate post-intervention | 3.94 (0.16) | 3.72 (0.18)
  6 months post-intervention | 4.10 (0.16) | 3.80 (0.18)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.2960, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in fruit & vegetable consumption scores from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.1519, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in fruit & vegetable consumption scores from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change in Proportion of Participants Engaging in Sufficient Levels of Physical Activity
Description: Change in proportion of participants engaging in sufficient levels of physical activity (PA) from baseline to immediate post-intervention and 6 months post-intervention. This measure assessed participants' frequency of engaging in both moderate and vigorous PA over the past month (>4 times a week, 2-4 times a week, about once a week, etc.). This measure was adapted to include relevant cultural examples of PA from the Dietary Approaches to Stop Hypertension 2 Brief Physical Activity Questionnaire (https://biolincc.nhlbi.nih.gov/media/studies/dashsodium/Forms_Manual.pdf?link_time=2018-11-13_18:06:05.776099). Both items used a 4-point response scale: 1) Rarely or Never; 2) Once a week; 3) 2-4 times a week; and 4) More than 4 times a week. Each 4-point scale for moderate PA and vigorous PA was weighted: 0=Rarely or Never; 1=Once a week; 2=2-4 times a week; and 4=More than 4 times a week. The weights were then summed and dichotomized as follows: ≥4 = sufficient PA and <4 = insufficient PA.
Time Frame: Baseline, immediate post-intervention, 6 months post-intervention
Population: Analysis includes only those with data on the relevant outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
Participants
  Baseline | 112 | 78
  Immediate post-intervention: number analyzed (Participants) | 171 | 111
  Immediate post-intervention | 108 | 63
  6 months post-intervention: number analyzed (Participants) | 171 | 116
  6 months post-intervention | 99 | 65
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Adjusted repeated measures generalized estimating equations (GEE) model; Test type: Superiority; p = 0.2824, Mantel Haenszel — The p-value above reflects results of between-arms analysis of change from baseline to immediate post-intervention. Analyses do not include imputed values; The model includes only the study arm and time interaction
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Adjusted repeated measures generalized estimating equations (GEE) model; Test type: Superiority; p = 0.7547, Mantel Haenszel — The p-value above reflects results of between-arms analysis of change from baseline to 6 months post-intervention. Analyses do not include imputed values; The model includes only the study arm and time interaction

8. Other Pre Specified Outcome: Change in Eating Habits Self-efficacy Score
Description: Change in eating habits self-efficacy from baseline to immediate post-intervention and 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' self-efficacy related to their ability to make healthy eating decisions in the face of real or perceived barriers (e.g. while at social events, while watching television, etc.). This 7-item measure was adapted from items in the original Weight Efficacy Life-Style (WEL) Questionnaire (Clark MM, Abrams DB, Niaura RS, et al. Self-efficacy in weight management. J Consult Clin Psychol. 1991;59(5):739-744). Each of the 7 items are measured via 3 response options ("Yes/Completely Sure"=2; "Maybe/Not Sure"=1; and "No/Not Sure at All"=0), giving a possible range of scores of 0-14, with higher scores indicating higher self-efficacy for making healthy eating decisions in spite of barriers.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: scale score
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
scale score
  Baseline | 10.97 (0.26) | 11.46 (0.28)
  Immediate post-intervention | 11.77 (0.28) | 11.92 (0.33)
  6 months post-intervention | 11.87 (0.28) | 11.62 (0.32)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.6928, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in eating self-efficacy scores from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.4947, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in eating self-efficacy scores from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

9. Other Pre Specified Outcome: Change in Physical Activity Self-efficacy
Description: Change in physical activity self-efficacy from baseline to immediate post-intervention and 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' self-efficacy for exercising in the face of real or perceived barriers (e.g., bad weather, exercising alone, etc.). This 9-item measure was adapted from the Self-Efficacy for Exercise (SEE) Scale (Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000;49(3):154-159. & Resnick B, Luisi D, Vogel A, Junaleepa P. Reliability and validity of the Self-Efficacy for Exercise and Outcome Expectations for Exercise Scales with minority older adults. J Nurs Measurement. 2004; 12(3):235-247.) Each of the 9 items are measured via 3 response options ("Yes/Completely Sure"=2; "Maybe/Not Sure"=1; and "No/Not Sure at All"=0), giving a possible range of scores of 0-18, with higher scores indicating higher self-efficacy.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: scale score
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
scale score
  Baseline | 13.64 (0.41) | 14.24 (0.45)
  Immediate post-intervention | 13.87 (0.44) | 14.72 (0.51)
  6 months post-intervention | 14.34 (0.44) | 13.57 (0.50)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.1539, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in physical activity self-efficacy scores from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.1878, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in physical activity self-efficacy scores from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Change in Perceived Family Support for Exercise and Dietary Habits
Description: Change in perceived family support for exercise and dietary habits from baseline to immediate post-intervention and 6 months post-intervention. This self-report measure was adapted to examine changes in perceived family support for engaging in healthy exercise and dietary habits. This measure consists of a 6-item scale adapted from: Gruber KJ. Social support for exercise and dietary habits among college students. Adolescence. 2008;43(171):557-575. Each of the 6 items are measured via 3 response options ("Often"=2; "Sometimes"=1; and "Never"=0), giving a possible range of scores of 0-12, with higher scores indicating higher perceived family support for exercising and eating healthier.
Time Frame: Baseline, Immediate post-intervention, 6 months post-intervention
Measure: Mean (Standard Error); unit: scale score
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
Number analyzed (Participants) | 212 | 166
scale score
  Baseline | 4.99 (0.25) | 5.50 (0.27)
  Immediate post-intervention | 6.66 (0.27) | 6.38 (0.31)
  6 months post-intervention | 6.48 (0.27) | 6.46 (0.31)
Statistical Analysis 1: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.4322, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in family support scale scores from baseline to immediate post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program vs Partnership for Improving Lifestyle Intervention Diabetes Prevention Program; Repeated measures regression model used all available participant data (no listwise deletion); Test type: Superiority; p = 0.9529, linear mixed effects regression — The p-value above reflects results of between-arms analysis of mean change in family support scale scores from baseline to 6 months post-intervention. Analyses do not include imputed values; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From enrollment to 1 year post-enrollment
Description: Study staff assessed presence of adverse events via regular contact with participants from both study arms throughout the duration of the study.
Arm/Group | Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program | Partnership for Improving Lifestyle Intervention Diabetes Prevention Program
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/167
Other Adverse Events (participants affected / at risk) | 0/213 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT03270436/Prot_SAP_000.pdf